CLINICAL TRIAL: NCT03567278
Title: Feasibility Trial on ACURATE™ Transapical Implantation in Patients With Severe Symptomatic Aortic Stenosis
Brief Title: Feasibility Trial on ACURATE™ Transapical Implantation in Patients With Severe Symptomatic Aortic Stenosis (2009-01)
Acronym: TA-FIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-01; DE/CA84/73-KL-30-09 (Other: Landesdirektion Sachsen - Freistaat Sachsen)
Record Dates: First submitted 2014-12-08; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-05

CONDITIONS: Aortic Stenosis Symptomatic
Keywords: Severe Symptomatic Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Medical Device Study
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACURATE TA™ (Experimental): Patients implanted with ACURATE TA™ Bioprosthesis
  Interventions: Device: ACURATE TA™

INTERVENTIONS:
Device: ACURATE TA™ — ACURATE TA™ Transapical Aortic Bioprosthesis is intended for subjects with severe symptomatic Aortic Stenosis and are considered high risk for surgical conventional Aortic Valve Replacement surgery.
  Other Names: ACURATE TA™ Transapical Aortic Bioprosthesis and Delivery System

SUMMARY:
Feasibility Trial on the ACURATE TA™ transapical implantation in patients presenting severe symptomatic aortic stenosis to collect human feasibility data pertaining to the safety and performance of the device.

DETAILED DESCRIPTION:
A single arm, prospective, multicenter, open trial up to 5 year follow-up with the SYMETIS ACURATE TA™ which is an aortic bioprosthesis for minimal invasive implantation via transapical access to treat patients with severe symptomatic aortic stenosis where conventional aortic valve replacement (AVR) via open heart surgery is considered to be associated with high surgical risk for evaluating the feasibility and performance of the implantation and the safety at 30-Day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 75 years;
* Additive EuroSCORE > 9 and/or STS > 9%;
* Severe symptomatic AS assessed by echocardiography, documented by a derived mean gradient > 40mmHg,and a native Aortic Valve Area (AVA) < 0.8 cm² or Aortic Valve Area Index (AVAI) < 0.6 cm²/m²;
* NYHA Functional Class > II;
* Aortic annulus (AAn) diameters between and including 21 mm up to 27 mm (21mm ≤ AAn ≤27mm) by transoesophageal echocardiography;
* Sinotubular junction (STJ) higher than 1,1times the native aortic annulus diameter (AAn) [STJ>1.1xAAn] AND STJ<45mm by transoesophageal echocardiography;
* Patient understands the implications of participating in the study and provides signed informed consent

Exclusion Criteria:

* Congenital unicuspid or bicuspid aortic valve;
* Severe eccentricity of calcification;
* Severe mitral regurgitation (> 2°);
* Pre-existing prosthetic heart valve in any position and /or prosthetic ring;
* Severe transapical access problem, non-reachable LV apex;
* Previous surgery of the LV using a patch, such as the Dor procedure;
* Presence of apical LV thrombus;
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation;
* Acute Myocardial Infarction (AMI) within 1 month prior to the procedure;
* PCI within 1 month prior to the procedure;
* Previous Transient Ischemic Accident (TIA) or stroke in the last 3 months;
* Untreated clinically significant CAD requiring revascularization;
* Hemodynamic instability: systolic pressure <90mmHg without afterload reduction, shock, need for inotropic support or intra-aortic balloon pump;
* Severe left ventricular dysfunction with a LV Ejection Fraction (LVEF) < 25% by echocardiography;
* Calcified pericardium;
* Septal hypertrophy;
* Primary Hypertrophic Obstructive Cardiomyopathy (HOCM);
* Active infection, endocarditis or pyrexia;
* Active peptic ulcer or Gastrointestinal (GI) bleeding within the past 3 months;
* Significant hepatic involvement (Child > B);
* Major lung disease (FEV < 0.8 or FEV1% < 30% of normal);
* Pulmonary hypertension;
* History of bleeding diathesis or coagulopathy;
* Hematologic disorder (WBC<3000mm3, Hb<9g/dL, platelet count <50000 cells/ mm3);
* Serum creatinine level greater than 3.0 mg/dL or chronic renal failure requiring dialysis;
* Neurological disease severely affecting ambulation or daily functioning, including dementia;
* Other procedure scheduled at the same time, whether surgery or percutaneous approach;
* Emergency procedure;
* Life expectancy < 12 months due to non-cardiac co-morbid conditions;
* Known hypersensitivity/contraindication to any study medication, contrast media, or nitinol;
* Currently participating in an investigational drug or another device study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety endpoint | 30 days
  Rate of Major Adverse Valve-Related Events (MAVRE) related to ACURATE

SECONDARY OUTCOMES:
Performance endpoint | Up to 24-hours post-procedure
  Stable ACURATE placement at intended site as assessed by angiography
Performance endpoint | Up to 24-hours post-procedure
  Adequate ACURATE device function as assessed by echocardiography
Mortality | 30 days, 60 days, 3 months, 6 months and 12 months
  Freedom from Death at follow-up
MAVRE at follow-up | discharge or 7 days, 3 months, 6 months and 12 months
  Rate of MAVRE at follow-up
MACCE or Major Adverse Cardiac and Cerebrovascular Event | 1 month, 3 months, 6 months and 12 months
  Rate of MACCE at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Mohr, Professor, Principal Investigator — Herzzentrum Leipzig GmbH
Locations (5):
- Germany (5):
  - Kerckhoff Klinik GmbH, Bad Nauheim
  - Universitätsklinikum Essen Westdeutsches Herzzentrum Essen, Essen
  - Universitätsklinikum Freiburg Herz- und Gefäßchirurgie, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf Klinik für Herz-und Gefäßchirurgie, Hamburg
  - Herzzentrum Leipzig GmbH, Leipzig

IPD SHARING:
Plan to Share IPD: No